CLINICAL TRIAL: NCT06318143
Title: mAnaging siCkle CELl disEase Through incReased AdopTion of hydroxyurEa in Nigeria
Acronym: ACCELERATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U01HL168084 (NIH)
Record Dates: First submitted 2024-02-20; First posted 2024-03-19 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-06

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (No Intervention): provision of information about task sharing
- TASSH (Experimental): replicable evidence-based task-sharing strategy,TAsk-Strengthening Strategy for Hemoglobinopathies (TASSH)
  Interventions: Behavioral: TASSH

INTERVENTIONS:
Behavioral: TASSH — Strategy for Hemoglobinopathies (TASSH) containing the essential components of i) Training healthcare workers/providers to be more patient-centered in clinical consultations, ii) Clinical reminders, and iii) Practice facilitation (TCP) known as (TASSH TCP) for SCD management (Figure 1A describes the components of the intervention).
  Arms: TASSH

SUMMARY:
Large knowledge gaps remain regarding strategies to promote the adoption of hydroxyurea (HU), particularly in sub-Saharan African countries including Nigeria, where more than 75% of annual sickle cell anemia births occur. The vast majority of people with SCD in Africa do not receive evidenced-based health care (e.g., newborn screening, health education, prophylaxis for infection, optimal nutrition and hydration, blood transfusion, transcranial Doppler screening, and HU therapy), despite its effectiveness in reducing SCD-related adverse outcomes and mortality. The use of HU in SSA is <1% among SCD patients. The investigators' preliminary findings indicate that provider-level barriers are significant and must be addressed to improve HU adoption. To address HU adoption, the investigators will use the NIH-funded study (e.g., Realizing Effectiveness Across Continents with Hydroxyurea (REACH) Clinical Trial (NCT01966731)) that developed an evidence-informed, clinical, practical, and easy-to-follow algorithm to 1) Screen patients for sickle cell disease (SCD), 2) Initiate HU treatment, and 3) Maintain HU dosage over time (SIM) for the improved management of SCD as our intervention. The Nigerian government released guidelines supporting the SIM intervention for HU adoption for improved SCD management, and HU is on the list of essential medicines for Nigeria. The investigators' implementation strategy for improving SCD management in Nigeria uses a practical and replicable evidence-based task-sharing strategy, TAsk-Strengthening Strategy for Hemoglobinopathies (TASSH), adopted from the TAsk-Strengthening Strategy for Hypertension control (TASSH) trials in Ghana and Nigeria containing the essential components of i) Training healthcare workers/providers to be more patient-centered in clinical consultations, ii) Clinical reminders, and iii) Practice facilitation (TCP) known as (TASSH TCP) for SCD management. Using a sequential exploratory mixed-methods study design, the investigators will conduct this study using the Exploration, Preparation, Implementation, and Sustainment (EPIS) framework in four sequential phases to assess the effectiveness of SIM adoption by providers in the context of the TASSH TCP implementation strategy in Nigeria.

DETAILED DESCRIPTION:
Aim 1: Using the EPIS framework as a guide, identify and characterize the capacity of 20 SPARC-NEt clinical sites to adopt SIM and adapt a tailored healthcare worker TASSH Training + Clinical reminders + Practice facilitation (TASSH TCP) for SCD management.

Aim 2: Evaluate in a cluster RCT, the effect of the TASSH TCP (experimental condition) vs. receipt of educational information only on TASSH TCP (control) on the adoption of SIM (primary outcome) across 20 SPARC-NEt clinical sites at 12 months. Hypothesis 1: The level of SIM adoption will be higher in the SPARC- NEt clinical sites randomized to the experimental condition than those in control.

Aim 3: Evaluate the mediators of SIM+TASSH TCP adoption, implementation fidelity, and sustainability across SPARC-NEt clinical sites at 12 and 24 months. Hypothesis 2: Inner organizational context, outer context, and implementation process will influence adoption, fidelity, and sustainability of SIM+TASSH TCP at clinical sites.

Impact: The study leverages the infrastructure of the SPARC-NEt (U01HL156942) of Nigeria to assess the adoption of HU among providers to improve SCD management in a manner that is scalable and sustainable across Nigeria and identify best practices for implementing HU therapy in resource constrained settings.

ELIGIBILITY:
Inclusion Criteria:

* SCD patients18 years older that have provided consent;
* Pediatric SCD patients aged 9 months to 17 years with an accompanying guardian and have provided informed consent or assent;
* Registration in the electronic medical records (EMR) database with clinical charts and received care at the local clinical sites or health facilities and not on HU therapy;
* Hb Genotype: SCD-SS, SCD-Sβo thal, SCD-SOArab (On a case by case basis, a severely affected person with SCD-SC may be offered HU therapy under a modified treatment protocol)

Exclusion Criteria:

* Any SCD patient not registered in the EMR database without informed consent or assent;
* Physically unable to participate in study activities;
* An SCD patient on HU

Min Age: 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Patient numbers - screening | 12 months
  The number of patients taking HU identified through screening
Patient numbers - proportion on HU | 12 months
  The proportion of patients that on HU based on the REACH Clinical Trial algorithm tailored for aged 9 months through adulthood using SPARCO HU Guidelines
Patient numbers - dosage | 12 months
  Proportion of patients who maintained HU dosage

SECONDARY OUTCOMES:
Mediators | 12 months and 24 months
  Secondary outcome measures are the mediators of SIM adoption and sustainability across the clinical sites at 12 and 24 months. The following measures will be used to assess the mediators of SIM via self-report. The mediators are based on the constructs of the EPIS including inner context characteristics of the clinics, intervention characteristics, and implementation process measures

CONTACTS AND LOCATIONS:
Locations (1):
- University Of Abuja Teaching Hospital, Abuja, Nigeria

REFERENCES:
- [Derived] Peprah E, Gyamfi J, Patena J, Kayalioglu H, Hameed T, Ogedegbe G, Do H, Ojji D, Adenikinju D, Ajaye Oba T, Nwegbu M, Isa H, Shedul G, Sopekan AY, Nnodu OE. An implementation trial to mAnage siCkle CELl disEase through incReased AdopTion of hydroxyurEa in Nigeria (ACCELERATE): Study protocol. PLoS One. 2025 Jan 8;20(1):e0311900. doi: 10.1371/journal.pone.0311900. eCollection 2025. PMID 39774400